CLINICAL TRIAL: NCT02437448
Title: Exhaled Breath Analysis by Secondary Electrospray Ionization - Mass Spectrometry (SESI-MS) in Patients With Pulmonary Fibrosis
Brief Title: Breath Analysis in Lung Fibrosis
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Collaborators: Swiss Federal Institute of Technology (Other); Swiss National Science Foundation (Other)
Responsible Party: Principal Investigator, Malcolm Kohler, Prof, University of Zurich
Other Study IDs: KEK-ZH-Nr. 2014-0573
Record Dates: First submitted 2015-04-28; First posted 2015-05-07 (Estimated); Last update posted 2020-10-05 (Actual); Status verified 2020-10

CONDITIONS: Idiopathic Lung Fibrosis; Idiopathic Pulmonary Fibrosis
Keywords: Mass spectrometry; Exhaled breath analysis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: None Retained — Exhaled breath
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Idiopathic lung fibrosis: 20 IPF patients
  Interventions: Other: No intervention
- Controls: 20 subjects with no apparent lung disease and normal lung function testing. Matched for gender, age and smoking history.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention

SUMMARY:
The aim of the study is to answer the question whether a disease specific profile of breath in patients with idiopathic lung fibrosis can be detected by an untargeted metabolomic study using exhaled breath analysis by mass spectrometry.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical symptoms consistent with IPF
2. Age 40 through 80 years
3. Diagnosis of UIP or IPF by HRCT and surgical lung biopsy as outlined in table 1. Only patients fulfilling the category "YES" will be included in the study.
4. Extent of fibrotic changes (honeycombing, reticular changes) greater than extent of emphysema on HRCT scan
5. No features supporting an alternative diagnosis

Exclusion Criteria:

1. Acute exacerbation within the last 6 weeks.
2. Any relevant lung disease other than pulmonary fibrosis.
3. Acute inflammatory disease (e.g. common cold) within the last 6 weeks.
4. Acute or chronic hepatic disease.
5. Renal failure or renal replacement therapy.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Confirmed diagnosis of idiopathic pulmonary fibrosis based on clinical, radiologic and/or pathologic data without evidence or suspicion of an alternative diagnosis that may contribute to their interstitial lung disease. Patients must fulfill all of the following criteria:
Sampling Method: Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2015-06; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
IPF-specific mass spectrometric profile of volatile organic compounds of exhaled breath analysis (markers of IPF in exhaled breath) | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Pulmonary Division, University Hospital of Zurich, Zurich, Switzerland

REFERENCES:
- [Derived] Gaugg MT, Engler A, Bregy L, Nussbaumer-Ochsner Y, Eiffert L, Bruderer T, Zenobi R, Sinues P, Kohler M. Molecular breath analysis supports altered amino acid metabolism in idiopathic pulmonary fibrosis. Respirology. 2019 May;24(5):437-444. doi: 10.1111/resp.13465. Epub 2019 Jan 25. PMID 30681243